CLINICAL TRIAL: NCT06905262
Title: Tumor Antigen Discovery for Innovative Cancer Immunotherapies in HCC: from Benchside to Bedside (HepAnt) - Study of the Role of the Metagenome in Head and Neck Tumors Using Omics Techniques - HeNomics
Brief Title: Tumor Antigen Discovery for Innovative Cancer Immunotherapies in HCC: from Benchside to Bedside (HepAnt)
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Other Study IDs: 57/22 oss (HepAnt)
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Tumor Antigen Discovery for Innovative Cancer Immunotherapies in HCC: From Benchside to Bedside (HepAnt) - Study of the Role of the Metagenome in Head and Neck Tumors Using Omics Techniques (HeNomics).

DETAILED DESCRIPTION:
The aim of this study is to:

* Analyze and compare the microbiota and the intestinal, salivary and intratumoral microbiome in patients with HCC, patients diagnosed with oncological pathology and in healthy subjects. The analysis of the mycobiota will be carried out by analyzing bacterial culture media, that of the microbiome by genomic analysis. The evaluation will be made by taking into account multiple taxonomic levels: phylum, class, order, family, genus and species.
* Identify tumor antigens (TuAs) with sequence homology with peptides derived from the microbiota/microbiome by bioinformatic analysis. The sequences of tumor antigens known from the literature (https://caped.icp.ucl.ac.be/Peptide/list) will be aligned with sequences derived from bacteria identified in the microbiota/microbiome of patients and healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of primary HCC and other oncological pathology (Pascale Institute) or diagnosis of oncological pathology (without any exclusions) from an accredited medical-clinical facility (Fortore Mountain Community).
* Age ≥18 years
* Ability to give signed informed consent that includes compliance with the requirements and constraints listed in the informed consent form (ICF) and in this protocol.
* In the case of paraffin-embedded samples obtained from the UOC of Pathological Anatomy and/or the Institute's Biological Bank, informed consent cannot be acquired, in accordance with the Provision of the Privacy Authority containing the requirements relating to the processing of special categories of data, pursuant to art. 21, paragraph 1 of Legislative Decree 10 August 2018, no. 101, published in the Official Journal - general series - no. 176 of 29/07/2019, point 5 "Provisions relating to the processing of personal data carried out for scientific research purposes (gen. aut. n. 9/2016)" HEALTHY SUBJECTS
* clinical history free from diagnosis of tumor or neoplastic pathology treated during life
* Age ≥80 years
* Ability to give signed informed consent that includes compliance with the requirements and constraints listed in the informed consent form (ICF) and in this protocol

Exclusion Criteria:

* Current pathologies requiring antibiotic therapy
* Diagnosis of pre-tumor pathology (in healthy subjects)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Patients with primary hepatocellular carcinoma attending the Institute for medical/surgical treatment (surgery, locoregional treatments, systemic pharmacological treatments). In addition, patients with a diagnosis of oncological pathology attending the Institute will be enrolled. With regard to the latter, this also includes patients who have already undergone surgery in the past and whose paraffin-coated tissues are preserved.
  * Healthy subjects over eighty years of age with a clinical history free from a diagnosis of tumor or neoplastic pathology treated during their life. The choice of these control subjects not matched by age to the patients is based on the rationale that they can be considered de facto "protected" from the tumor pathology. Consequently, they represent the true negative control of the study.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-01-02 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Identification and classification of the numerical variation | approximately 16 months
  Identification and classification of the numerical variation (appearance or disappearance) of bacterial species and/or their representativeness (percentage of the total) in the intestinal, salivary and intratumoral microbiota/microbiome of the two groups of enrolled subjects.
Identification and classification of the different number and identity of antigens | approximately 16 months
  Identification and classification of the different number and identity of antigens predicted by the bacterial species present in the intestinal, salivary and intratumoral microbiota/microbiome of the two groups of enrolled subjects.
Identification and classification of the number and identity of TuAs | approximately 16 months
  Identification and classification of the number and identity of TuAs that share sequence homology with peptides derived from bacteria that are components of the intestinal, salivary and intratumoral microbiota/microbiome of the two groups of enrolled subjects.

SECONDARY OUTCOMES:
Identification of the percentage of memory CD8+ T lymphocytes | approximately 16 months
  - Identification of the percentage of memory CD8+ T lymphocytes in the two groups of enrolled subjects showing cross-reactivity against TuAs and epitopes derived from bacteria that are components of the intestinal, salivary and intratumoral microbiota/microbiome.
Identification and classification of numerical variation | approximately 16 months
  Identification and classification of the numerical variation (appearance or disappearance) and/or their representativeness (percentage of the total) of the TCR sequences of CD8+ T cells in the two groups of enrolled subjects cross-reactive with TuAs and epitopes derived from bacteria that are components of the intestinal, salivary and intratumoral microbiota/microbiome.

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Buonaguro, Principal Investigator — IRCCS I.N.T. "G. Pascale"
Locations (1):
- Istituto Nazionale Tumori di Napoli - IRCCS - Fondazione G. Pascale, Napoli, Italy